CLINICAL TRIAL: NCT05278728
Title: Phase IIa Study of Nimotuzumab Plus Irinotecan as Second-line Treatment in Metastatic Colorectal Cancer With Wild Type K-ras
Brief Title: Phase IIa Study of Nimotuzumab to Treat Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT-CRC-T
Record Dates: First submitted 2015-08-18; First posted 2022-03-14 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer
Keywords: nimotuzumab; colorectal cancer; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — nimotuzumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nimotuzumab and Irinotecan (Experimental): Nimotuzumab： 200, 400, 600 or 800mg weekly until progression or AEs Irinotecan：180mg/m2 d1, Q2w until progression or AEs or maximum 6 cycles
  Interventions: Drug: Nimotuzumab; Drug: Irinotecan

INTERVENTIONS:
Drug: Nimotuzumab — 200,400,600 or 800mg weekly until progression or AEs
Drug: Irinotecan — 180mg/m2 d1, Q2w until progression or AEs or maximum 6 cycles

SUMMARY:
Nimotuzumab is an IgG1 humanized monoclonal antibody that recognized an epitope located in the extra cellular domain of the human epidermal growth factor receptor (EGFR). Clinical efficacy has been shown in adult with head and neck cancer. The study assessed the safety, and efficacy of the combination of Nimotuzumab administered concomitantly with chemotherapy in patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
Nimotuzumab and Irinotecan will be administered to the patient until disease progression or development of toxicity preclude further treatment. Irinotecan will be administered once every 14 days, the dosage is 180mg/m2; Nimotuzumab treatment be divided 3 levels: 200mg/w, 400mg/w, 600mg/w, weekly. The patients'blood test and liver and renal function tests will be monitored weekly, a physical exam and reassessment of the tumor will be performed and every 6 weeks, when the total result is the CR or PR, the result of the 6th and the 12th week should be compared.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed before performing any of the study's specific procedures.
* ECOG performance status 0-2.
* Age > 18，both genders.
* Metastatic colorectal cancer confirmed by pathology, or locally advanced unresectable colorectal cancer, or postoperative recurrence and metastasis colorectal cancer
* Disease progression after receiving oxaliplatin ± fluorouracil in first-line treatment
* At least 1 measurable lesions ,( longest diameter≥ 1 cm by spiral computed tomography (CT) scan or MRI)
* Life expectancy more than 3 months.
* K-ras is wild type
* Use of an effective contraceptive method for patients of both sexes when there is a risk of conception and/or pregnancy.
* Liver metastasis, lesions smaller than 50% of the liver; Lung metastasis, lesions smaller than 30% of the lung
* Haemoglobin≥90g/L , granulocyte≥1.5×109/L ,WBC ≥3×109/L, platelet count≥100×109/L
* TBIL≤ 1.5 x ULN ,ALK≤ 2.5 x ULN or ≤ 5ULN（Liver metastasis），AST and ALT≤ 2.5 x ULN or ≤ 5ULN（Liver metastasis）,Creatinine ≤ 1.5 x ULN
* No brain metastasis

Exclusion Criteria:

* Previous radiotherapy at lesions within three months
* Other first line chemo-agents treatment except oxaliplatin ± fluorouracil
* Received other anti EGFR monoclonal antibody treatment
* Complete or incomplete intestinal obstruction
* Participation in other interventional clinical trials within 1 month
* Psychiatric disease affected cognitive ability, including brain metastasis
* Peripheral neuropathy lesion is more than I stage.
* History of serious allergic or allergy
* Pregnant or breast-feeding women
* Patients with the history of Serious lung or hear disease
* Other malignant tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-07; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The rate of grade 3/4 toxicity | 3 months
  The rate of grade 3/4 toxicity, defined as the proportion or frequency of patients who experience toxicity reactions that are classified as grade 3 or grade 4 according to CTCAE v5.0.

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 3 months
  Rate of dose-limiting toxicities (DLTs) after infusion of nimotuzumab. The highest dose at which 0 or 1 DLT occurs in 6 DLT-evaluable subjects will be declared the maximum tolerated dose (MTD).
The complete response rate | 3 months
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: Complete Response (CR), defined as the disappearance of all target lesions.
The partial response rate | 3 months
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: Partial Response (PR), defined as at least a 30% decrease in the sum of the longest diameter of target lesions.
The disease control rate | 3 months
  Disease control rate (DCR), including complete response (CR) and partial response (PR) and stable disease(SD). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: CR, disappearance of all target lesions; PR, at least a 30% decrease in the sum of the longest diameter of target lesions. SD, neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (PD, defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions).

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Department of GI Oncology,Peking University, School of Oncology, Beijing Cancer Hospital & Institute
Locations (2):
- China (2):
  - China People's Liberation Army (PLA)81 Hospital, Nanjing, Jiangsu
  - Peking University, School of Oncology, Beijing Cancer Hospital & Institute, Beijing